CLINICAL TRIAL: NCT01873872
Title: Evaluation of Probiotics and the Development of Clostridium Difficile Associated Diarrhea in Patients Receiving Antibiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Vincent's East, Birmingham, Alabama (Other)
Collaborators: Master Supplements, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROBIOTIC
Record Dates: First submitted 2013-06-05; First posted 2013-06-10 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2013-06

CONDITIONS: Development of Clostridium Difficile Associated Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Theralac probiotic (Active Comparator)
  Interventions: Dietary Supplement: Theralac probiotic
- Culturelle probiotic (Active Comparator)
  Interventions: Dietary Supplement: Culturelle probiotic
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Theralac probiotic
  Arms: Theralac probiotic
Dietary Supplement: Culturelle probiotic
  Arms: Culturelle probiotic
Other: placebo
  Arms: Placebo

SUMMARY:
We have designed this study to measure the effect of normal flora supplementation, using available probiotics, on the incidence of Clostridium difficile-associated diarrhea

in a population of general inpatients who are receiving antibiotics.

DETAILED DESCRIPTION:
General medical-surgical patients in a community hospital who are receiving antibiotics, and who agree to participate, will be given one of two different probiotics, or placebo. Data will be gathered during their hospitalization, and at one and three months following hospital discharge. We expect to see a lower incidence of Clostridium difficile-associated diarrhea in the probiotic groups when compared to the placebo group. We will also be looking for differences between the effects of the two probiotics, which differ in strain types and number of colony forming units per dose.

ELIGIBILITY:
Inclusion Criteria: Any hospitalized patient who is age 19 or older and receiving antibiotics.

-

Exclusion Criteria:

* Feeding tube in place
* Pregnancy
* Milk or soy allergy
* Sensitivity to lactose
* Immunocompromised defined as:

  1. Absolute neutrophil count (ANC) ≤ 500 cells/mm3
  2. HIV
  3. Cancer patient receiving chemotherapy or radiation therapy
  4. Immune deficiency
  5. Post organ transplant

Participants will be withdrawn from the study if they develop any of the exclusion criteria during the hospitalization.

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Development of Clostridium difficile associated diarrhea in patients receiving antibiotics | Up to six months

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Phillips, Pharm.D, Principal Investigator — St. Vincent's East; Walter Ross, MD, Principal Investigator — St. Vincent's East; Mark Middlebrooks, MD, Principal Investigator — St. Vincent's East; Lee Wimberly, MD, Principal Investigator — St. Vincent's East; Linda Adams, RPh, Principal Investigator — St. Vincent's East; Carrie Castleberry, RN, Principal Investigator — St. Vincent's East
Locations (1):
- St. Vincent's East, Birmingham, Alabama, United States